CLINICAL TRIAL: NCT06261710
Title: Intrapartum Ultrasound in Labor: Sonography Only, Few Internal Examinations
Acronym: SOFIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Larry Hinkson (Other)
Responsible Party: Sponsor-Investigator, Larry Hinkson, Principal Investigator, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EA2_253_23
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Labor Complication
Keywords: Chorioamnionitis; Sonography
MeSH Terms: conditions — Obstetric Labor Complications; Chorioamnionitis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonography Only (Experimental): The use of ultrasound parameters to asses the progress of labour from admission to delivery. Namely, Angle of Progression, Head Perineum Distance, Midline Angle and Cervix Dilatation at 3-4 hour intervals until delivery.
  Interventions: Other: Sonography in labour
- Traditional (No Intervention): The traditional use of internal vaginal examination to assess cervix dilatation, fetal head position, station and orientation within the pelvis during the course of labour as routinely performed every 3-4 hours in labour and until delivery.

INTERVENTIONS:
Other: Sonography in labour — Using intrapartum sonography parameters in labour
  Arms: Sonography Only

SUMMARY:
This is a prospective, randomized trial to determine whether the use of sonographic parameters during labor results in less intrapartum infection compared to traditional invasive examination. Other secondary outcomes include maternal satisfaction and overall birth outcomes.

DETAILED DESCRIPTION:
It is a prospective, randomized trial to determine whether the use of sonographic parameters during childbirth results in less intrapartum infection compared to traditional invasive examination. Intrapartum non-invasive ultrasound has been established and validated as a method of assessing labor progress. Guidelines from international societies recommend the use of ultrasound to monitor labor and support decision-making during delivery. Despite its reproducibility and reliability, there is no comprehensive work to date demonstrating the potential benefit in reducing clinical chorioamnionitis compared to traditional invasive vaginal examination. With this in mind, the investigators set out to analyze the clinical benefit of using ultrasound alone using established non-invasive, intrapartum, translabial parameters (Angle of Progression, Head Perineum Distance, Midline Angle, Cervix Dilatation) to monitor birth outcomes compared to traditional invasive vaginal examinations.

Primary Outcome is the incidence of clinical chorioamnionitis. Secondary Outcome measures include mode of delivery and neonatal outcomes such as neonatal admission.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of at least 18 years of age with a singleton in the cephalic position
* Spontaneous onset of labor; births after induction of labor with otherwise suitable inclusion and exclusion criteria are also permitted.

Exclusion Criteria:

* Emergency situations such as maternal or fetal bleeding
* Indication for urgent delivery by caesarean section
* Pathological cardiotocogram
* non-cephalic positions
* under 18 years of age
* women giving birth who are unable to give consent

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 356 (Estimated)
Dates: Start 2024-02-27 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Maternal Fever Incidence | In the course of labour from admission until delivery in 3-4 hour intervals
  Percentage. Incidence of Fever >37.8°C measured with a thermometer in patients within the group
Maternal Tachycardia Incidence | In the course of labour from admission until delivery in 3-4 hour intervals
  Percentage. Incidence of >100 beats per minute as maternal pulse measurement in patients within the group
Maternal Leucocytosis | In the course of labour from admission until delivery in 6 hour intervals
  Percentage. Incidence of maternal leucocytosis (white blood cell count >15,000 leukocytes per microliter of blood) in patients within the group
Uterine tenderness | In the course of labour from admission until delivery 3-4 hour intervals
  Percentage. The incidence of uterine tenderness on palpation during the course of labour in patients within the group
Fetal Tachycardia | In the course of labour from admission until delivery
  Percentage.The incidence of fetal tachycardia (>160 beats per minute) on continuous Cardiotocographic Monitoring in patients within the group
Foul-smelling amniotic fluid | In the course of labour from admission until delivery
  Percentage . The incidence of foul-smelling amniotic fluid on clinical examination in patients with in the group

SECONDARY OUTCOMES:
Average age | Upon admission for delivery
  Number (years) measured per patient and the average within the group.
Maternal weight | Upon admission for delivery
  Number (kilograms) measured per patient and the average within the group.
Maternal height | Upon admission for delivery
  Number (centimetres) measured per patient and the average within the group.
Completed weeks of pregnancy | Upon admission for delivery
  Number (weeks) measured per patient and the average within the group.
Previous pregnancy | Upon admission for delivery
  Number measured per patient and the average within the group.
Incidence of Vaginal Examinations | In the course of labour until delivery
  Percentage. The number of vaginal examinations performed in labour on average per patient within the group.
Incidence of Caesarean section | In the course of labour until delivery
  Percentage.The incidence of Caesarean section (No. of Cesareans as a percentage of the Group total)
Incidence of Instrumental Delivery | In the course of labour until delivery
  Percentage.The incidence of instrumental deliveries (No. of instrumental deliveries as a percentage of the total in the group)
Incidence of estimated blood loss >1000 ml | In the course of labour until delivery and up to 24 hours postpartum
  Percentage.The incidence of estimated blood loss >1000 millilitres (No. of cases as a percentage of the total in the group)
Incidence of antibiotics usage | In the course of labour until delivery and up to 24 hours postpartum
  Percentage.The incidence of antibiotic use (No. of cases as a percentage of the total in the group)
Incidence of Neonatal Admission | Up to 6 weeks postpartum
  Percentage. The incidence of neonatal admission in patients within the groups
Neonatal weight | Up to 30 Minutes after birth
  Number. Gramms measures on weighing on a scale
Maternal Satisfaction Scores | On admission and after delivery
  Linkert scores. Questionnaire on maternal views on the use of examination in labour. (Linkert scores from 1-6 with increasing scale)

OTHER OUTCOMES:
Incidence of Chorioamnionitis on Placenta Histologie | After delivery up to 6 weeks postpartum
  Percentage. Incidence of Histological Chorioamnionitis on histological examination of the placenta in patients within the group

CONTACTS AND LOCATIONS:
Overall Officials: Larry Hinkson, FRCOG, Principal Investigator — Charité University Hospital Department of Obstetrics
Locations (1):
- Charité University Hospital, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tita AT, Andrews WW. Diagnosis and management of clinical chorioamnionitis. Clin Perinatol. 2010 Jun;37(2):339-54. doi: 10.1016/j.clp.2010.02.003. PMID 20569811
- [Background] Ghi T, Eggebo T, Lees C, Kalache K, Rozenberg P, Youssef A, Salomon LJ, Tutschek B. ISUOG Practice Guidelines: intrapartum ultrasound. Ultrasound Obstet Gynecol. 2018 Jul;52(1):128-139. doi: 10.1002/uog.19072. PMID 29974596